CLINICAL TRIAL: NCT04887584
Title: Identifying the Role of Pulses in a Healthful Diet: Metabolomic Signatures of Dietary Pulses and Their Benefits on Cardiometabolic Risk Factors
Brief Title: Pulse Biomarker Discovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: FL115
Record Dates: First submitted 2021-05-10; First posted 2021-05-14 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Body Weight
Keywords: Dietary pulses; Urine biomarkers; Microbiome; Short chain fatty acids; Plasma biomarkers; Fecal biomarkers; Beans; Lentils; Controlled feeding; Intervention; Chickpeas; Metabolomics
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Masking Description: Unblinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Group 1 (Experimental): Order of treatments:
  A: Control diet B: Low pulse diet C: High pulse diet
  Interventions: Other: Control diet; Other: Low Pulse diet; Other: High Pulse diet
- Group 2 (Experimental): Order of treatments:
  A: Control diet C: High pulse diet B: Low pulse diet
  Interventions: Other: Control diet; Other: Low Pulse diet; Other: High Pulse diet
- Group 3 (Experimental): Order of treatments:
  B: Low pulse diet A: Control diet C: High pulse diet
  Interventions: Other: Control diet; Other: Low Pulse diet; Other: High Pulse diet
- Group 4 (Experimental): Order of treatments:
  B: Low pulse diet C: High pulse diet A: Control diet
  Interventions: Other: Control diet; Other: Low Pulse diet; Other: High Pulse diet
- Group 5 (Experimental): Order of treatments:
  C: High pulse diet A: Control diet B: Low pulse diet
  Interventions: Other: Control diet; Other: Low Pulse diet; Other: High Pulse diet
- Group 6 (Experimental): Order of treatments:
  C: High pulse diet B: Low pulse diet A: Control diet
  Interventions: Other: Control diet; Other: Low Pulse diet; Other: High Pulse diet

INTERVENTIONS:
Other: Control diet — The control Typical American Diet (TAD) diet pattern will mimic the level of intake of fruits, vegetables, whole grains, added sugars, saturated fats and sodium in the general U.S. population. This diet will feature no servings of pulses per day.
Other: Low Pulse diet — The Low Pulse diet will be designed based on the TAD with substitution of pulses for lean meat and grains. This diet will feature 0.2 cups of pulses per day at 2,000 kilocalories (kcals).
Other: High Pulse diet — The High Pulse diet will be designed based on the TAD with substitution of pulses for lean meat and grains. This diet will feature 1.5 cups of pulses per day at 2,000 kilocalories (kcals).

SUMMARY:
Dietary pulses, including beans, chickpeas, and lentils, are high in soluble fiber with potential benefits to human health: Pulses are moderate energy density foods, low in fat and high in dietary protein, fiber, vitamins and minerals. Moderate pulse consumption is associated with improvements in glycemic control and reduced risk of cardiovascular disease, obesity and type 2 diabetes. Measuring pulse consumption in humans is difficult, due to limitations in current methods for dietary assessment which are largely based on dietary recalls that are subject to reporting bias. Robust tools for pulse intake assessment are needed, and biomarkers of dietary pulse intake are one approach to solve this problem. The goal of this human feeding study is evaluate the presence of biomarkers of dietary pulses in human subjects.

DETAILED DESCRIPTION:
Dietary pulses, including beans, chickpeas, and lentils, are high in soluble fiber with potential benefits to human health: Pulses are moderate energy density foods, low in fat and high in dietary protein, fiber, vitamins and minerals. Moderate pulse consumption is associated with improvements in glycemic control and reduced risk of cardiovascular disease, obesity and type 2 diabetes. However, only 5% of the U.S. population currently meet recommended fiber intakes. As pulses are an excellent source of fiber, increasing their levels in the American diet could lead to demonstrable health benefits in the population, including positive influences on glucose regulation. Additionally, pulse impacts on the gut microbiome may be responsible for reported health benefits. While diet has direct impacts on health, these effects can be mediated by the microbiome, and dietary fiber is a key determinant of this interaction. The fermentation of soluble fiber by specific microbial species lead to the production of short chain fatty acids (SCFAs) including propionate and butyrate which are positively associated with insulin sensitivity. In general, elevated colonic SCFA production is associated with improved glucose regulation, appetite modulation, and immune system modulation.

The overall goal of this research is to evaluate how pulse digestion and microbial fermentation influence the circulating and excreted metabolome. To achieve this goal, a randomized controlled feeding study including one week of control, low pulse and high pulse diet will be provided to participants. Metabolomics will be used to identify biomarkers or signatures for pulse enriched diets in urine and plasma. In addition, researchers will investigate dietary pulse related changes in the microbiome community and short chain fatty acid production in fecal samples.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) 18-30 kg/m2
* Willingness to provide urine and stool and have blood drawn

Exclusion Criteria:

* Active participation in another research study
* Tested positive for severe acute respiratory syndrome (SARS) Coronavirus (COV)-2 within the past 10 days
* Been in close contact with a SARS COV-2 positive person within the past 14 days
* Unwillingness to consume pulses or pulse-related products
* Fasting glucose ≥120 mg/dL
* Fasting triglyceride ≥400 mg/dL
* LDL-cholesterol ≥160 mg/dL
* Blood Pressure (BP): Systolic BP ≥140 mmHg or Diastolic BP ≥90 mmHg
* Current use of dietary supplements and/or unwillingness to cease intake of dietary supplements

  * Vegan or vegetarian lifestyle or any other dietary restrictions that would interfere with consuming the intervention foods and beverages (including dietary intolerances, allergies and sensitivities)
  * Unwillingness to consume intervention foods and beverages
  * Engage in

    * More than moderate drinking (> 1 drink serving per day for women or >2 drink servings per day for men).
    * Binge drinking (4 drinks within two hours).
  * Excessive intake of caffeine containing products (excessive defined as ≥ 400mg/day)
  * Diagnosis of disordered eating or eating disorder
  * Recent diagnosis of any of the following or measurement on screening lab tests

    * Anemia (hemoglobin <11.7g/dL)
    * Abnormal liver function
    * Liver Enzymes that are >200% of upper limit (alanine aminotransferase (ALT) upper limit is 43 U/L or aspartate aminotransferase (AST) upper limit is 54 U/L)
  * History of any of the following

    * Gastric bypass surgery
    * Inflammatory bowel disease (IBD) or other GI conditions that would interfere with consuming the intervention foods
    * Active cancer in the past three years excluding squamous or basal cell carcinomas of the skin that have been handled medically by local excision
    * Other serious medical conditions
  * Recent dental work or have conditions of the oral cavity that would interfere with consuming the intervention foods and beverages
  * Long term use of antibiotics
  * Taking any over the counter or prescribed medication for any of the following

    * Elevated lipids or glucose
    * High blood pressure
    * Weight loss
  * Are pregnant, planning to become pregnant within the duration of the study or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2023-11-07 (Actual)

PRIMARY OUTCOMES:
Change in urine metabolomics profile | Day 14, 28, and 42; fasting and post prandial 0.5hr, 2hr, 3hr, 6hr, 12hr and 24hr
  Urine metabolites will be measured by gas chromatography mass spectrometry (GCMS) before and after consumption of control, low pulse or high pulse diets.
Change in plasma metabolomics profile | Day 14, 28, and 42; fasting and post prandial 0.5hr, 2hr, 3hr and 6hr
  Plasma metabolites will be measured by gas chromatography mass spectrometry (GCMS) before and after consumption of control, low pulse or high pulse diets.

SECONDARY OUTCOMES:
Change in fecal microbiome community | Day 7, 14, 21, 28, 35, 42
  DNA of colonic microbiome will be measured before and after each diet exposure.
Change in fecal short chain fatty acids | Day 7, 14, 21, 28, 35, 42
  Acetate, propionate and butyrate will be measured by GCMS before and after each diet exposure.
Change in fecal bile acids | Day 7, 14, 21, 28, 35, 42
  Bile acids will be measured by GCMS before and after each diet exposure.
Change in plasma short-chain fatty acids | Day 14, 28, and 42; fasting and post prandial 0.5hr, 2hr, 3hr and 6hr
  Plasma acetate, propionate and butyrate will be measured by GCMS before and after consumption of control, low pulse or high pulse diets.
Change in pro-inflammatory cytokines | Day 14, 28, and 42; fasting and post prandial 0.5hr, 2hr, 3hr and 6hr
  Cytokines including tumor necrosis factor alpha (TNF-a), interleukin (IL)-1, IL-6 and interferon-gamma will be measured in plasma using multiplex assays.
Change in anti-inflammatory cytokines | Day 14, 28, and 42; fasting and post prandial 0.5hr, 2hr, 3hr and 6hr
  Cytokines including interleukin (IL)-1 receptor antagonist, IL-4, IL-10, IL-11, and IL-13 will be measured in plasma using multiplex assays.

CONTACTS AND LOCATIONS:
Overall Officials: Brian J Bennett, PhD, Principal Investigator — USDA ARS Western Human Nutrition Research Center
Locations (1):
- USDA ARS Western Human Nutrition Research Center, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCrory MA, Hamaker BR, Lovejoy JC, Eichelsdoerfer PE. Pulse consumption, satiety, and weight management. Adv Nutr. 2010 Nov;1(1):17-30. doi: 10.3945/an.110.1006. Epub 2010 Nov 16. PMID 22043448
- [Background] Margier M, George S, Hafnaoui N, Remond D, Nowicki M, Du Chaffaut L, Amiot MJ, Reboul E. Nutritional Composition and Bioactive Content of Legumes: Characterization of Pulses Frequently Consumed in France and Effect of the Cooking Method. Nutrients. 2018 Nov 4;10(11):1668. doi: 10.3390/nu10111668. PMID 30400385
- [Background] Mudryj AN, Yu N, Aukema HM. Nutritional and health benefits of pulses. Appl Physiol Nutr Metab. 2014 Nov;39(11):1197-204. doi: 10.1139/apnm-2013-0557. Epub 2014 Jun 13. PMID 25061763
- [Background] Jenkins DJ, Kendall CW, Augustin LS, Mitchell S, Sahye-Pudaruth S, Blanco Mejia S, Chiavaroli L, Mirrahimi A, Ireland C, Bashyam B, Vidgen E, de Souza RJ, Sievenpiper JL, Coveney J, Leiter LA, Josse RG. Effect of legumes as part of a low glycemic index diet on glycemic control and cardiovascular risk factors in type 2 diabetes mellitus: a randomized controlled trial. Arch Intern Med. 2012 Nov 26;172(21):1653-60. doi: 10.1001/2013.jamainternmed.70. PMID 23089999
- [Background] Anderson JW, Baird P, Davis RH Jr, Ferreri S, Knudtson M, Koraym A, Waters V, Williams CL. Health benefits of dietary fiber. Nutr Rev. 2009 Apr;67(4):188-205. doi: 10.1111/j.1753-4887.2009.00189.x. PMID 19335713
- [Background] Threapleton DE, Greenwood DC, Evans CE, Cleghorn CL, Nykjaer C, Woodhead C, Cade JE, Gale CP, Burley VJ. Dietary fibre intake and risk of cardiovascular disease: systematic review and meta-analysis. BMJ. 2013 Dec 19;347:f6879. doi: 10.1136/bmj.f6879. PMID 24355537
- [Background] Yao B, Fang H, Xu W, Yan Y, Xu H, Liu Y, Mo M, Zhang H, Zhao Y. Dietary fiber intake and risk of type 2 diabetes: a dose-response analysis of prospective studies. Eur J Epidemiol. 2014 Feb;29(2):79-88. doi: 10.1007/s10654-013-9876-x. Epub 2014 Jan 5. PMID 24389767
- [Background] Quagliani D, Felt-Gunderson P. Closing America's Fiber Intake Gap: Communication Strategies From a Food and Fiber Summit. Am J Lifestyle Med. 2016 Jul 7;11(1):80-85. doi: 10.1177/1559827615588079. eCollection 2017 Jan-Feb. PMID 30202317
- [Background] Makki K, Deehan EC, Walter J, Backhed F. The Impact of Dietary Fiber on Gut Microbiota in Host Health and Disease. Cell Host Microbe. 2018 Jun 13;23(6):705-715. doi: 10.1016/j.chom.2018.05.012. PMID 29902436
- [Background] Muller M, Hernandez MAG, Goossens GH, Reijnders D, Holst JJ, Jocken JWE, van Eijk H, Canfora EE, Blaak EE. Circulating but not faecal short-chain fatty acids are related to insulin sensitivity, lipolysis and GLP-1 concentrations in humans. Sci Rep. 2019 Aug 29;9(1):12515. doi: 10.1038/s41598-019-48775-0. PMID 31467327
- [Background] Wrzosek L, Miquel S, Noordine ML, Bouet S, Joncquel Chevalier-Curt M, Robert V, Philippe C, Bridonneau C, Cherbuy C, Robbe-Masselot C, Langella P, Thomas M. Bacteroides thetaiotaomicron and Faecalibacterium prausnitzii influence the production of mucus glycans and the development of goblet cells in the colonic epithelium of a gnotobiotic model rodent. BMC Biol. 2013 May 21;11:61. doi: 10.1186/1741-7007-11-61. PMID 23692866
- [Background] McRorie JW Jr, McKeown NM. Understanding the Physics of Functional Fibers in the Gastrointestinal Tract: An Evidence-Based Approach to Resolving Enduring Misconceptions about Insoluble and Soluble Fiber. J Acad Nutr Diet. 2017 Feb;117(2):251-264. doi: 10.1016/j.jand.2016.09.021. Epub 2016 Nov 15. PMID 27863994
- [Background] Parada Venegas D, De la Fuente MK, Landskron G, Gonzalez MJ, Quera R, Dijkstra G, Harmsen HJM, Faber KN, Hermoso MA. Short Chain Fatty Acids (SCFAs)-Mediated Gut Epithelial and Immune Regulation and Its Relevance for Inflammatory Bowel Diseases. Front Immunol. 2019 Mar 11;10:277. doi: 10.3389/fimmu.2019.00277. eCollection 2019. PMID 30915065
- [Background] Garcia-Mantrana I, Selma-Royo M, Alcantara C, Collado MC. Shifts on Gut Microbiota Associated to Mediterranean Diet Adherence and Specific Dietary Intakes on General Adult Population. Front Microbiol. 2018 May 7;9:890. doi: 10.3389/fmicb.2018.00890. eCollection 2018. PMID 29867803
- [Background] Gibson RS, Charrondiere UR, Bell W. Measurement Errors in Dietary Assessment Using Self-Reported 24-Hour Recalls in Low-Income Countries and Strategies for Their Prevention. Adv Nutr. 2017 Nov 15;8(6):980-991. doi: 10.3945/an.117.016980. Print 2017 Nov. PMID 29141979
- [Background] Corrigendum for McCullough et al. Metabolomic markers of healthy dietary patterns in US postmenopausal women. Am J Clin Nutr 2019;109:1439-51. Am J Clin Nutr. 2020 Mar 1;111(3):728. doi: 10.1093/ajcn/nqz235. No abstract available. PMID 32115661
- [Background] Ross AB, Bourgeois A, Macharia HN, Kochhar S, Jebb SA, Brownlee IA, Seal CJ. Plasma alkylresorcinols as a biomarker of whole-grain food consumption in a large population: results from the WHOLEheart Intervention Study. Am J Clin Nutr. 2012 Jan;95(1):204-11. doi: 10.3945/ajcn.110.008508. Epub 2011 Dec 14. PMID 22170369
- [Background] Brennan L, Hu FB. Metabolomics-Based Dietary Biomarkers in Nutritional Epidemiology-Current Status and Future Opportunities. Mol Nutr Food Res. 2019 Jan;63(1):e1701064. doi: 10.1002/mnfr.201701064. Epub 2018 May 28. PMID 29688616
- [Background] Madrid-Gambin F, Llorach R, Vazquez-Fresno R, Urpi-Sarda M, Almanza-Aguilera E, Garcia-Aloy M, Estruch R, Corella D, Andres-Lacueva C. Urinary 1H Nuclear Magnetic Resonance Metabolomic Fingerprinting Reveals Biomarkers of Pulse Consumption Related to Energy-Metabolism Modulation in a Subcohort from the PREDIMED study. J Proteome Res. 2017 Apr 7;16(4):1483-1491. doi: 10.1021/acs.jproteome.6b00860. Epub 2017 Mar 16. PMID 28067528
- [Background] Mifflin MD, St Jeor ST, Hill LA, Scott BJ, Daugherty SA, Koh YO. A new predictive equation for resting energy expenditure in healthy individuals. Am J Clin Nutr. 1990 Feb;51(2):241-7. doi: 10.1093/ajcn/51.2.241. PMID 2305711